CLINICAL TRIAL: NCT04237935
Title: Replication of the PLATO Antiplatelet Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-PLATO
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Antiplatelet
MeSH Terms: interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clopidogrel 75 mg: Reference group
  Interventions: Drug: Clopidogrel 75mg
- Ticagrelor 90 mg: Exposure group
  Interventions: Drug: Ticagrelor 90mg

INTERVENTIONS:
Drug: Ticagrelor 90mg — Ticagrelor 90 mg dispensing claim is used as the exposure group
  Groups: Ticagrelor 90 mg
Drug: Clopidogrel 75mg — Clopidogrel 75 mg dispensing claim is used as the reference group
  Groups: Clopidogrel 75 mg

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Please see: https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

Market availability of ticagrelor in the U.S. started on 2011-07-20.

* For Marketscan: 2011-07-20 to 2017-12-31 (end of data availability).
* For Optum: 2011-07-20 to 2019-03-31 (end of data availability).

Inclusion Criteria:

* 1-4 ALL REQUIRED

  * 1. Hospitalized for potential ST-segment elevation or non-ST-segment elevation ACS, with onset during the previous 24 hours, documented by cardiac ischemic symptoms due to atherosclerosis of ≥10 minutes' duration at rest
  * 2. ≥18 years of age
  * 3. Not pregnant. Urinary and/or blood pregnancy tests are to be performed in women of child-bearing potential and repeated at least every 6 months. Women of child-bearing potential must be using ≥2 forms of reliable contraception, including one barrier method.
  * 4. With informed consent 1-4 AND 5A OR 5B
* 5A. ≥2 of the following:

  * 1. ST-segment changes on ECG indicating ischemia. ST-segment depression or transient elevation ≥ 1 mm in two or more 2 contiguous leads"
  * 2. Positive biomarker indicating myocardial necrosis. Troponin I or T or CK-MB greater than the upper limit of normal
  * 3. One of the following:

    1. ≥60 y of age
    2. Previous MI or CABG
    3. CAD with ≥50% stenosis in ≥2 vessels
    4. Previous ischemic stroke, TIA (hospital-based diagnosis), carotid stenosis (≥50%), or cerebral revascularization
    5. Diabetes mellitus
    6. Peripheral artery disease
    7. Chronic renal dysfunction
* OR
* 5B. Persistent ST-segment elevation ≥1 mm (not known to be preexisting or due to a coexisting disorder) in ≥2 contiguous leads or new LBBB plus primary PCI planned.

Exclusion Criteria:

* Drug related

  * 1. Contraindication to clopidogrel or other reason that study drug should not be administered (eg, hypersensitivity, moderate or severe liver disease, active bleeding or bleeding history, major surgery within 30 days)"
  * 2. Oral anticoagulation therapy that cannot be stopped
  * 3. Fibrinolytic therapy planned or within the previous 24 h
  * 4. Concomitant oral or IV therapy with strong CYP3A inhibitors (ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, grapefruit juice N1 L/d), CYP3A substrates with narrow therapeutic indices (cyclosporine, quinidine), or strong CYP3A inducers (rifampin/rifampicin, phenytoin, carbamazepine)
* Treatment related

  * 1. Index event is an acute complication of PCI
  * 2. PCI after index event and before first study dose
* Medical

  * 1. Increased risk of bradycardiac events
  * 2. Dialysis required
  * 3. Known clinically important thrombocytopenia
  * 4. Known clinically important anemia
  * 5. Any other condition that may put the patient at risk or influence study results in the investigators' opinion (eg, cardiogenic shock, severe hemodynamic instability, active cancer)
* General

  * 1. Participant in another investigational drug or device study within 30 days
  * 2. Pregnancy or lactation
  * 3. Any condition that increases the risk for noncompliance or being lost to follow-up
  * 4. Involvement in the planning or conduct of the study
  * 5. Previous enrollment or randomization in this study

Ages: 18 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, cohort study design comparing ticagrelor 90mg twice daily to clopidogrel 75mg daily. The patients will be required to have continuous enrollment during the baseline period of 180 days before initiation of ticagrelor 90mg or the comparator drug (cohort entry date). Follow-up for the outcome (3P-MACE), begins the day after drug initiation.
Sampling Method: Non-Probability Sample
Enrollment: 27960 (Actual)
Dates: Start 2019-09-22 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Relative hazard of 3-P MACE (composite outcome of Stroke, MI, and Mortality) | Through study completion (a median of 163-219 days)
  Relative hazard of 3-point major adverse cardiovascular events (MACE), i.e., non-fatal myocardial infarction, non-fatal stroke, or all-cause/CV mortality- Please refer to uploaded protocol for full definition due to size limitations.

SECONDARY OUTCOMES:
Relative hazard of Hospital admission for MI | Through study completion (a median of 163-219 days)
  Relative hazard of Hospital admission for MI - Please refer to uploaded protocol for full definition due to size limitations.
Relative hazard of Hospital admission for stroke | Through study completion (a median of 163-219 days)
  Relative hazard of Hospital admission for stroke - Please refer to uploaded protocol for full definition due to size limitations.
Relative hazard of All-cause mortality/CV mortality | Through study completion (a median of 163-219 days)
  Relative hazard of All-cause mortality/CV mortality- Please refer to uploaded protocol for full definition due to size limitations.

OTHER OUTCOMES:
Relative hazard of Major bleeding (Control outcome) | Through study completion (a median of 163-219 days)
  Relative hazard of Major bleeding (Control outcome) - Please refer to uploaded protocol for full definition due to size limitations.
Relative hazard of Pneumonia (Control outcome) | Through study completion (a median of 163-219 days)
  Relative hazard of Pneumonia (Control outcome) - Please refer to uploaded protocol for full definition due to size limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham And Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Franklin JM, Patorno E, Desai RJ, Glynn RJ, Martin D, Quinto K, Pawar A, Bessette LG, Lee H, Garry EM, Gautam N, Schneeweiss S. Emulating Randomized Clinical Trials With Nonrandomized Real-World Evidence Studies: First Results From the RCT DUPLICATE Initiative. Circulation. 2021 Mar 9;143(10):1002-1013. doi: 10.1161/CIRCULATIONAHA.120.051718. Epub 2020 Dec 17. PMID 33327727

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/35/NCT04237935/Prot_SAP_000.pdf